CLINICAL TRIAL: NCT06554080
Title: Survival and Success Rates of External- and Internal- Connection Dental Implants Placed Within the United Kingdom Armed Forces.
Status: Active, not recruiting | Type: Observational
Sponsor: Defence Primary Health Care, UK (Other Government)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 2303/MODREC/24
Record Dates: First submitted 2024-05-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant Failed; Tooth Loss; Implant Complication
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platform-matched: UK Armed Forces patients who had platform-switched implants (Nobel Brånemark or NobelSpeedy Groovy) placed at DCRD between the period of 01 Jan 2017 and 31 Dec 2023.
  Interventions: Procedure: Platform-matched implant placement
- Platform-switched: UK Armed Forces patients who had platform-switched implants (NobelParallel or NobelActive) placed at DCRD between the period of 01 Jan 2017 and 31 Dec 2023.
  Interventions: Procedure: Platform-switched implant placement

INTERVENTIONS:
Procedure: Platform-switched implant placement — NobelParallel or NobelActive implants placed
  Groups: Platform-switched
Procedure: Platform-matched implant placement — Nobel Brånemark, NobelSpeedy Groovy implants placed
  Groups: Platform-matched

SUMMARY:
This is a retrospective cohort study that evaluates the survival (Outcome 1) of dental implant systems (external connection (Cohort 1) and internal connection (Cohort 2) and the effectiveness of maintaining crestal bone levels (Outcome 2), placed within United Kingdom Armed Forces personnel. The secondary objectives include: assessment of block bone grafting on outcome, assessment of restoration (bridge vs crown on outcome) and assessment of placement technique (immediate, early, delayed placement). Inclusion criteria: all military patients that received dental implants since 2014-2024. Exclusion criteria: military patients that have not received radiographic review or follow-up of the dental implant or who have left service or have a follow-up that is less than 12-months post placement of the dental implant..

DETAILED DESCRIPTION:
Dental care to the United Kingdom Armed Forces (UKAF) is provided by Defence Primary Healthcare (DPHC) Dental, which incorporates a Managed Clinical Network (MCN) to co-ordinate and treat complex restorative cases referred by general dental practitioners (GDPs), with a central hub at the DCRD. The DCRD routinely employs dental implants within patients' rehabilitative treatment pathways.

Nobel Biocare are the sole provider of dental implants to DPHC with three-systems (Nobel Speedy Groovy, Nobel Active and Nobel Parallel) routinely employed. Of the three systems, Nobel Speedy Groovy have been in use for over 20-years, employing an external hexagon prosthet-ic connection (EH). With EH, the microbiological junction lies at the vertical junction of the abutment and implant (Platform-Matched (P-M)). Subsequently, a 1mm zone of inflammation occurs around this junction with associated crestal bone loss. The establishment of crestal bone levels at the first thread of the implant was within the parameters of implant success. In contrast, Nobel Active and Parallel systems employ an internal conical connection (CC) that facilitates a platform-switching (P-S) approach to restoration of the implant. The platform switching concept aims to move the microbiological junction to the horizontal coronal surface of the implant, away from the implant/ alveolar junction, with the aim of preserving vertical crestal bone to the full height of the implant. This study aims to evaluate whether platform-switching influences dental implant survival (primary outcome) and radiographic bone levels (secondary outcome).

The study aims to account for the following factors on the outcome measures: dental implant pathway protocol (immediately-, early-, delayed- or late-placement protocols post extraction), bone grafting (to facilitate implant provision) either undertaken either prior to- or during- implant placement (block grafting, sinus floor elevation, augmentation at time of placement) and restoration type (crown, bridge, over-denture support).

ELIGIBILITY:
Inclusion Criteria:

* • Military patients who had dental implants placed at DCRD between the period of 01 Jan 2017 and 31 Dec 2023.

  * Patients over the age of 18 (female) and 19 (male, to allow for recommended lower age limits for implant placement due to facial growth).
  * Healthy and medically compromised patients (diabetes mellitus type-2 (DM2), systemic steroid usage, immune-supressed patients, smoking habits).
  * Implants placed with concomitant grafting or in a site where socket-preservation procedure completed.
  * Patients with periodontal health as well as history of periodontal disease.
  * Dental Implant types to include Nobel Biocare; Parallel, Active, Branemark and SpeedyGroovy.
  * Implants with immediate, early, delayed and late implant placement pathways.
  * Implants restored with single unit and multi-unit fixed prostheses.
  * Minimum of 12-month follow-up data available.
  * Pre-operative long cone periapical (LCPA) radiographs available to view at surgical placement, implant restoration and follow-up (12-month).

Exclusion Criteria:

* • Implants placed outside of DPHC.

  * Implants placed in sites where a block-grafts or sinus floor elevation procedure completed.
  * Implants supporting removable prostheses.
  * Implants placed prior to- or after- closure of trial period.
  * Patients under the age of 18 (female) and 19 (male).
  * No follow-up LCPA.
  * Patients that died before pathway/ follow-up was completed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: UK Armed Forces
Sampling Method: Non-Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Dental Implant Survival (presence of implant at point of review) | Minimum time frame for inclusion is 12 months
  Null hypothesis: No difference in dental implant survival between the 2 cohorts (Platform-Matched vs Platform-Switched dental implant/ abutment interfaces). This is a binary outcome of either implant still present or implant absent at time of review.

SECONDARY OUTCOMES:
Dental Implant Crestal Bone Levels | Minimum time frame for inclusion is 12 months
  Null hypothesis: There is no difference in the crestal bone levels between the 2 cohorts (Platform-Matched vs Platform-Switched dental implant/ abutment interfaces). This outcome is measured radiographically using a software programme to determine changes in bone levels. Outcome is measured in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Defence Centre of Rehabiliative Dentistry, Aldershot, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No